CLINICAL TRIAL: NCT01023919
Title: Assessment of Surface Coverage of Polymer-based Sirolimus-eluting Stent( Cypher ) or Polymer-free Paclitaxel-eluting Stent (YinYi )in Diabetes Mellitus and Non- Diabetes Mellitus Patients by Optical Coherence Tomography
Brief Title: Assessment of Surface Coverage of Two Types of Drug-eluting Stent in Diabetes Mellitus and Non-Diabetes Mellitus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in enrolling the required number of participants has made it impractical to proceed with the trial.
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yu Bo, Prof, Harbin Medical University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HMUOCT-DM vs NDM-2
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus
Keywords: Optical coherence tomography; Drug eluting stent; Coronary Artery Disease; Diabetes Mellitus
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group B: (Active Comparator): Coronary artery disease without diabetes mellitus
  Interventions: Device: Device: Polymer-based sirolimus-eluting stent(Cypher stent ) and Polymer-free paclitaxel-eluting stent (YinYi stent)
- Group A: (Active Comparator): Coronary artery disease with diabetes mellitus
  Interventions: Device: Device: Polymer-based sirolimus-eluting stent(Cypher stent ) and Polymer-free paclitaxel-eluting stent (YinYi stent)

INTERVENTIONS:
Device: Device: Polymer-based sirolimus-eluting stent(Cypher stent ) and Polymer-free paclitaxel-eluting stent (YinYi stent) — Cypher stent or YinYi stent randomly implanted in coronary artery disease

SUMMARY:
Diabetic patients are prone to a diffuse and rapidly progressive form of atherosclerosis. Both clinical and angiographic outcomes following percutaneous coronary intervention (PCI) are poor in patients with DM compared with those without DM. Autopsy study has shown delayed neointimal healing with inadequate endothelialization and persistent stent surface ﬁbrin deposition after DES implantation in DM patients. This might partially contribute to the high risk of late stent thrombosis.

YINYI Polymer-Free paclitaxel stent is a domestic new type stent with bare metal base with micro porous surface. However, limited data is available in vivo about the surface coverage after stent implantation in DM patients because of lack of sensitive imaging modalities. Optical coherence tomography (OCT) is an optical analogue of intravascular ultrasound（IVUS）that allows high-resolution tomographic intravascular imaging. Furthermore, several studies have demonstrated the feasibility of OCT to quantitatively evaluate the surface coverage and stent conditions in the follow up after PCI .

Therefore, the aim of this study was to analyze the surface coverage and late malapposition after two types of DES implantation in DM patients compared with non-DM patients by using OCT and IVUS

DETAILED DESCRIPTION:
Diabetic patients are prone to a diffuse and rapidly progressive form of atherosclerosis. Both clinical and angiographic outcomes following percutaneous coronary intervention (PCI) are poor in patients with DM compared with those without DM. Autopsy study has shown delayed neointimal healing with inadequate endothelialization and persistent stent surface ﬁbrin deposition after DES implantation in DM patients. This might partially contribute to the high risk of late stent thrombosis.

YINYI Polymer-Free paclitaxel stent is a domestic new type stent with bare metal base with micro porous surface. However, limited data is available in vivo about the surface coverage after stent implantation in DM patients because of lack of sensitive imaging modalities. Optical coherence tomography (OCT) is an optical analogue of intravascular ultrasound（IVUS）that allows high-resolution tomographic intravascular imaging.

Therefore, the aim of this study was to analyze the surface coverage and late malapposition after two types of DES implantation in DM patients compared with non-DM patients by using OCT and IVUS

ELIGIBILITY:
Inclusion Criteria

General Inclusion Criteria：

1. Age : 18-75Y
2. Patients diagnosed as type 2 DM or non-DM.

Angiographic Inclusion Criteria：

1. Patients were considered eligible if they have one significant (>70%) angiographic stenosis lesions in native coronary vessel by CAG.
2. Each target is de novo lesion that can be treated with 1-2 stents.
3. Reference vessel diameter of 2.5 to 4.0 mm.

Exclusion Criteria

General Exclusion Criteria：

1. ST-segment elevation myocardial infarction within 7 days prior to the index procedure.
2. Life expectancy <12 months due to another medical condition.
3. Contraindication to antiplatelet therapy or a history of hypersensitivity to sirolimus and paclitaxel or structurally related compounds.
4. Creatinine level more than 2.0mg/dL or ESRD.
5. Severe hepatic dysfunction (more than 3 times normal reference values).
6. Planned surgery procedure≤12 months post-index procedure.
7. Known allergy to stainless steel.
8. Female of childbearing potential with a positive pregnancy test within 7 days before the index procedure, or lactating, or intends to become pregnant during the 12 months post index procedure.
9. Patient is not clinically appropriate for OCT evaluation in the opinion of investigator.

Angiographic Exclusion Criteria：

1. Study lesion is ostial in location (within 3.0 mm of vessel origin).
2. Study lesion involving arterial segments with highly tortuous anatomy.
3. Complex lesion morphologies (bifurcation needs two stents technique, left main lesion, chronic obstructive occlusion, severe thrombus, heavy calcification).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To investigate the difference of surface coverage pattern between diabetic patients and non-diabetic patients after DES (Cypher stent or YINYI stent)implantation | 6 months
  To investigate the difference of surface coverage pattern between diabetic patients and non-diabetic patients after DES (Cypher stent or YINYI stent)implantation

SECONDARY OUTCOMES:
To investigate the difference of surface coverage pattern between diabetic patients and non-diabetic patients after DES (Cypher stent or YINYI stent) implantation | 12 months
  To investigate the difference of surface coverage pattern between diabetic patients and non-diabetic patients after DES (Cypher stent or YINYI stent) implantation
To investigate the incidence of malapposition between diabetic patients and non-diabetic patients after DES (Cypher stent or YINYI stent) implantation | 6 months
  To investigate the incidence of malapposition between diabetic patients and non-diabetic patients after DES (Cypher stent or YINYI stent) implantation
To investigate the incidence of malapposition between diabetic patients and non-diabetic patients after DES (Cypher stent or YINYI stent) implantation | 12 months
  To investigate the incidence of malapposition between diabetic patients and non-diabetic patients after DES (Cypher stent or YINYI stent) implantation
To investigate the differences of surface coverage pattern，the incidence of malapposition and in-stent thrombosis between Cypher stent and YINYI in diabetic patients | 6 and 12 months.
  To investigate the differences of surface coverage pattern，the incidence of malapposition and in-stent thrombosis between Cypher stent and YINYI in diabetic patients
To investigate the differences of surface coverage pattern，malapposition and the incidence of thrombosis between Cypher stent and YINYI in non-diabetic patients | 6 and 12 months.
  To investigate the differences of surface coverage pattern，malapposition and the incidence of thrombosis between Cypher stent and YINYI in non-diabetic patients

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yu, MD,PhD, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University
Locations (1):
- The second Affiliated Hospital of Harbin Medical University, Harbin, Heilong Jiang, China